CLINICAL TRIAL: NCT02083965
Title: A Randomized, Open-Label, Crossover Study to Evaluate the Pharmacokinetics of 2 Vial Strengths of Recombinant Factor VIII Fc Fusion Protein (rFVIIIFc; BIIB031) in Previously Treated Subjects With Severe Hemophilia A
Brief Title: Pharmacokinetics of rFVIIIFc at Two Vial Strengths
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioverativ Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 997HA307; 2013-003013-18 (EudraCT Number)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2017-05

CONDITIONS: Severe Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII-Fc fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rFVIIIFc 1000 / 3000 PK Assessment (Experimental): A single intravenous (IV) injection of rFVIIIFc 50 IU/kg at a strength of 1000 IU/vial followed by a single IV injection of rFVIIIFc 50 IU/kg at a strength of 3000 IU/vial.
  Following the PK assessment, participants will receive either an episodic (on-demand) regimen with doses between 20 and 50 IU/kg based on the severity of the bleeding episode, or 1 of 2 prophylactic regimens: 50 IU/kg every 3 to 5 days or 65 IU/kg weekly. Participants will be allowed to switch from one regimen to another if approved by the Investigator.
  Interventions: Biological: rFVIIIFc
- rFVIIIFc 3000 / 1000 PK Assessment (Experimental): A single IV injection of rFVIIIFc 50 IU/kg at a strength of 3000 IU/vial followed by a single IV injection of rFVIIIFc 50 IU/kg at a strength of 1000 IU/vial.
  Following the PK assessment, participants will receive either an episodic (on-demand) regimen with doses between 20 and 50 IU/kg based on the severity of the bleeding episode, or 1 of 2 prophylactic regimens: 50 IU/kg every 3 to 5 days or 65 IU/kg weekly. Participants will be allowed to switch from one regimen to another if approved by the Investigator.
  Interventions: Biological: rFVIIIFc

INTERVENTIONS:
Biological: rFVIIIFc — Administered as specified in the treatment arm.
  Other Names: Eloctate; antihemophilic factor [recombinant] FC fusion protein; recombinant coagulation factor VIII Fc fusion protein; efmoroctocog alfa; BIIB031; Elocta

SUMMARY:
The primary objective of the study is to characterize the pharmacokinetics (PK) of rFVIIIFc administered at vial strengths of 1000 and 3000 IU in subjects with severe hemophilia A. The secondary objective of the study is to evaluate the safety of rFVIIIFc beyond the PK assessment for up to 6 months for a continued treatment period.

DETAILED DESCRIPTION:
This is a randomized, open-label, crossover study during which each participant receives a single injection of rFVIIIFc from 2 different vial concentrations (PK assessment). After the PK assessment, participants are provided with rFVIIIFc for either prophylactic or episodic (on-demand) treatment for up to 6 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Have severe hemophilia A
* Previously treated subject, defined as having at least 150 documented prior exposure days to any recombinant and/or plasma-derived FVIII and/or cryoprecipitate products (other than any use of rFVIIIFc- study drug or commercial product) at Day 1. Fresh frozen plasma treatment must not be considered in the count for documented exposure days.
* No history of a positive inhibitor test or clinical signs of decreased response to FVIII administrations. Family history of inhibitors will not exclude subjects.
* No measurable inhibitor activity using the Nijmegen-modified Bethesda assay at Screening.
* Platelet count ≥100,000 platelets/μL at screening
* CD4 lymphocytes >200 mm3 if known as HIV antibody positive at screening.
* Viral load of <400 copies/mL if known HIV antibody positive at screening.

Key Exclusion Criteria:

* Subject is at high risk of bleeding during the 5-day period between the first and second injections for PK analyses, as per Investigator discretion.
* Previous treatment with rFVIIIFc as study drug or commercial product.
* Other coagulation disorder(s) in addition to hemophilia A.
* History of hypersensitivity or anaphylaxis associated with any FVIII or IV immunoglobulin administration.
* Currently taking (or likely to require during the study) acetylsalicylic acid (ASA), except for low-dose ASA as prophylaxis (other nonsteroidal anti-inflammatory drugs are permitted).
* Concurrent systemic treatment with immunosuppressive drugs within 12 weeks prior to Day 1. Exceptions to this include: ribavirin for treatment of hepatitis C virus (HCV), and/or systemic steroids (a total of 2 courses of pulse treatments lasting no more than 7 days at a dose of ≤1 mg/kg within 12 weeks prior to Day 1) and/or inhaled steroids.

NOTE: Other protocol-defined inclusion/exclusion Criteria May Apply

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Bioverativ Therapeutics Inc.
Locations (8):
- United States (3):
  - Research Site, Los Angeles, California
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
- Australia (2):
  - Research Site, Herston
  - Research Site, Perth
- United Kingdom (3):
  - Research Site, Basingstoke
  - Research Site, Cambridge
  - Research Site, London

RESULTS

PARTICIPANT FLOW:
Groups:
- rFVIIIFc 1000 / 3000: Following a minimum 4-day washout, participants received a single injection 50 IU/kg at strength of 1000 IU/vial of rFVIIIFc (on Injection 1 Day 1) with 96 hours of pharmacokinetic (PK) assessments followed by a minimum of a 5-day washout prior to a second single injection of rFVIIIFc 50 IU/kg at strength of 3000 IU/vial (on Injection 2 Day 1) with 96 hours of PK assessments.
  After completing the PK assessment, all participants began 1 of 3 continued treatment regimens for up to 6 months:
  1. A prophylaxis regimen at a starting dose of 50 IU/kg of rFVIIIFc given every 3 to 5 days; further dose and interval adjustments were based on the Investigator's discretion as needed to prevent or treat bleeding.
  2. A prophylaxis regimen of 65 IU/kg administered every 7 days was considered for appropriate subjects who were selected based on the opinion of the Investigator.
  3. An episodic (on-demand) treatment with rFVIIIFc at 20 to 50 IU/kg, depending on the severity of the bleeding episode.
- rFVIIIFc 3000 / 1000: Following the minimum 4-day washout, participants received a single injection 50 IU/kg at strength of 3000 IU/vial of rFVIIIFc (on Injection 1 Day 1) with 96 hours of PK assessments followed by a minimum of a 5-day washout prior to a second single injection of rFVIIIFc 50 IU/kg at a strength of 1000 IU/vial (on Injection 2 Day 1) with 96 hours of PK assessments.
  After completing the PK assessment, all participants began 1 of 3 continued treatment regimens for up to 6 months:
  1. A prophylaxis regimen at a starting dose of 50 IU/kg of rFVIIIFc given every 3 to 5 days; further dose and interval adjustments were based on the Investigator's discretion as needed to prevent or treat bleeding.
  2. A prophylaxis regimen of 65 IU/kg administered every 7 days was considered for appropriate subjects who were selected based on the opinion of the Investigator.
  3. An episodic (on-demand) treatment with rFVIIIFc at 20 to 50 IU/kg, depending on the severity of the bleeding episode.
Period: PK Period 1
Arm/Group | rFVIIIFc 1000 / 3000 | rFVIIIFc 3000 / 1000
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | rFVIIIFc 1000 / 3000 | rFVIIIFc 3000 / 1000
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: PK Period 2
Arm/Group | rFVIIIFc 1000 / 3000 | rFVIIIFc 3000 / 1000
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0
Period: Treatment Period
Arm/Group | rFVIIIFc 1000 / 3000 | rFVIIIFc 3000 / 1000
Started | 10 | 8 (1 participant completed PK period 1 and 2, then chose to withdraw and did not enter treatment period)
Completed | 9 | 8
Not Completed | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- rFVIIIFc 1000 / 3000: Following the minimum 4-day washout, participants received a single injection 50 IU/kg at strength of 1000 IU/vial of rFVIIIFc (on Injection 1 Day 1) with 96 hours of PK assessments followed by a minimum of a 5-day washout prior to a second single injection of rFVIIIFc 50 IU/kg at a strength of 3000 IU/vial (on Injection 2 Day 1) with 96 hours of PK assessments.
  After completing the PK assessment, all participants began 1 of 3 continued treatment regimens for up to 6 months:
  1. A prophylaxis regimen at a starting dose of 50 IU/kg of rFVIIIFc given every 3 to 5 days; further dose and interval adjustments were based on the Investigator's discretion as needed to prevent or treat bleeding.
  2. A prophylaxis regimen of 65 IU/kg administered every 7 days was considered for appropriate subjects who were selected based on the opinion of the Investigator.
  3. An episodic (on-demand) treatment with rFVIIIFc at 20 to 50 IU/kg, depending on the severity of the bleeding episode.
- Total: Total of all reporting groups
Arm/Group | rFVIIIFc 1000 / 3000 | rFVIIIFc 3000 / 1000 | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (12.45) | 30.9 (19.76) | 26.7 (16.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) as Measured by Activated Partial Thromboplastin Time (aPTT) Clotting Assay
Description: Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞).
Time Frame: Predose, 0.5 hour (+-5 minutes); 1 hour and 6 hours (+-10 minutes); and 24, 48, 72, and 96 hours (+-60 minutes) after each injection
Population: The Pharmacokinetic Analysis Set is defined as all eligible participants who received at least one dose of rFVIIIFc and had sufficient PK data points to calculate at least one of the PK parameters of interest from either the aPTT clotting assay or the two-stage chromogenic clotting assay.
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Groups:
- rFVIIIFc 1000 IU: a single injection of rFVIIIFc 50 IU/kg at a strength of 1000 IU/vial
- rFVIIIFc 3000 IU: a single injection of rFVIIIFc 50 IU/kg at a strength of 3000 IU/vial
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
IU*h/dL | 2888.9 [2440.0 to 3420.5] | 2646.3 [2149.8 to 3257.5]

2. Primary Outcome: Incremental Recovery (IR, K Value) as Estimated From the FVIII Activity Data Measured by aPTT Clotting Assay
Description: The rise in FVIII activity in IU/dL per unit dose administered in IU/kg (IR, K value), as estimated from the FVIII activity data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 18 | 18
IU/dL | 2.33 [2.182 to 2.487] | 2.412 [2.169 to 2.682]

3. Secondary Outcome: Maximum Activity (Cmax) as Measured by the aPTT Clotting Assay
Description: Maximum measured concentration of rFVIIIFc.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 18 | 18
IU/dL | 122.2 [113.77 to 131.25] | 129.08 [114.62 to 145.37]

4. Secondary Outcome: Half-life (t½) as Measured by aPTT Clotting Assay
Description: Time required for the concentration of the drug to reach half of its original value.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
hours | 18.28 [16.10 to 20.75] | 17.49 [15.22 to 20.10]

5. Secondary Outcome: Clearance (CL) as Measured by the aPTT Clotting Assay
Description: The measure of the efficiency of the body to remove the drug and the unit is the volume of the plasma or blood cleared of drug per unit time.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
mL/h/kg | 1.807 [1.534 to 2.128] | 2.016 [1.642 to 2.476]

6. Secondary Outcome: Volume of Distribution at Steady State (Vss) as Measured by the aPTT Clotting Assay
Description: The apparent volume of distribution at steady state. (Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
mL/kg | 47.00 [43.87 to 50.35] | 48.65 [44.83 to 52.79]

7. Secondary Outcome: Mean Residence Time (MRT) as Measured by the aPTT Clotting Assay
Description: The average time at which the number of absorbed molecules reside in the body, after single-dose administration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
hours | 26.01 [22.49 to 30.08] | 24.13 [20.46 to 28.46]

8. Secondary Outcome: Time of Cmax (Tmax) as Measured by aPTT Clotting Assay
Description: Time at which maximum activity (Cmax) is observed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Groups:
- rFVIIIFc 3000 IU: rFVIIIFc single injection 50 IU/kg at a strength of 3000 IU/vial
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 18 | 18
hours | 0.66 [0.55 to 0.79] | 0.58 [0.51 to 0.67]

9. Secondary Outcome: Area Under the Curve to the Last Measurable Time Point (AUClast) as Measured by aPTT Clotting Assay
Description: Area under the plasma concentration time-curve from zero to the last measured concentration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
IU*h/dL | 2792.5 [2378.5 to 3278.6] | 2562.2 [2100.8 to 3125.0]

10. Secondary Outcome: Terminal Exponential Rate Constant (Lambda Z) as Measured by aPTT Clotting Assay
Description: First order rate constant associated with the terminal portion of the curve (lambda z) .
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: 1/h
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
1/h | 0.03792 [0.03340 to 0.04304] | 0.03963 [0.03449 to 0.04554]

11. Secondary Outcome: Percentage of AUCinf From the Last Data Point to Infinity (AUCext) as Measured by aPTT Clotting Assay
Description: Percentage of AUCinf extrapolated from the last data point to infinity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of AUCinf
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
percentage of AUCinf | 2.561 [1.703 to 3.852] | 2.279 [1.505 to 3.45]

12. Secondary Outcome: Dose Normalized Area Under the Curve (DNAUC) as Measured by aPTT Clotting Assay
Description: Dose normalized area under the FVIII activity-time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL per IU/kg
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
IU*h/dL per IU/kg | 55.35 [47.00 to 65.18] | 49.6 [40.4 to 60.9]

13. Secondary Outcome: Terminal Exponential Volume of Distribution (Vz) as Measured by aPTT
Description: The theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
mL/kg | 47.65 [43.73 to 51.93] | 50.87 [45.56 to 56.8]

14. Secondary Outcome: AUCinf as Estimated From the FVIII Activity Data as Measured by Two-Stage Chromogenic Clotting Assay
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 15 | 16
IU*h/dL | 2649.0 [2230.2 to 3146.5] | 2628.0 [2206.2 to 3130.5]

15. Secondary Outcome: IR, K Value as Measured by Two-Stage Chromogenic Clotting Assay
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL per IU/kg
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
IU/dL per IU/kg | 2.535 [2.245 to 2.862] | 2.287 [2.010 to 2.601]

16. Secondary Outcome: Cmax as Measured by Two-Stage Chromogenic Clotting Assay
Description: Maximum measured concentration of rFVIIIFc.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/dL
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
IU/dL | 132.61 [116.85 to 150.50] | 122.29 [106.80 to 140.03]

17. Secondary Outcome: t½ as Measured by Two-Stage Chromogenic Clotting Assay
Description: Time required for the concentration of the drug to reach half of its original value.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 15 | 16
hours | 18.58 [16.35 to 21.12] | 19.10 [16.44 to 22.19]

18. Secondary Outcome: CL as Measured by Two-Stage Chromogenic Clotting Assay
Description: as for outcome 5
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mL/h/kg
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 15 | 16
mL/h/kg | 1.962 [1.665 to 2.311] | 2.006 [1.720 to 2.339]

19. Secondary Outcome: Vss as Measured by Two-Stage Chromogenic Clotting Assay
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Groups:
- rFVIIIFc 3000 IU: a single injection of rFVIIIFc 50 IU/kg at a strength of 1000 IU/vial
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 15 | 16
mL/kg | 47.41 [43.01 to 52.26] | 51.27 [44.65 to 58.88]

20. Secondary Outcome: MRT as Measured by Two-Stage Chromogenic Clotting Assay
Description: The average time at which the number of absorbed molecules reside in the body, after single-dose administration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 15 | 16
hours | 24.17 [21.16 to 27.60] | 25.56 [22.15 to 29.50]

21. Secondary Outcome: Tmax as Measured by Two-Stage Chromogenic Clotting Assay
Description: Time at which maximum activity (Cmax) is observed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 17 | 18
hours | 0.61 [0.51 to 0.71] | 0.61 [0.52 to 0.72]

22. Secondary Outcome: AUClast as Measured by Two-Stage Chromogenic Clotting Assay
Description: Area under the plasma concentration time-curve from zero to the last measured concentration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 15 | 16
IU*h/dL | 2555.4 [2166.7 to 3013.9] | 2520.5 [2124.4 to 2990.5]

23. Secondary Outcome: Lambda Z as Measured by Two-Stage Chromogenic Clotting Assay
Description: First order rate constant associated with the terminal portion of the curve (lambda z).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: 1/h
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 15 | 16
1/h | 0.03730 [0.03282 to 0.04239] | 0.03629 [0.03124 to 0.04216]

24. Secondary Outcome: AUCext as Measured by Two-Stage Chromogenic Clotting Assay
Description: Percentage of AUCinf extrapolated from the last data point to infinity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of AUCinf
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 15 | 16
percentage of AUCinf | 2.923 [2.106 to 4.057] | 2.965 [1.890 to 4.650]

25. Secondary Outcome: DNAUC as Measured by Two-Stage Chromogenic Clotting Assay
Description: Dose normalized area under the FVIII activity-time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU*h/dL per IU/kg
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 15 | 16
IU*h/dL per IU/kg | 50.97 [43.27 to 60.05] | 49.85 [42.75 to 58.13]

26. Secondary Outcome: Vz as Measured by Two-Stage Chromogenic Clotting Assay
Description: as for outcome 13
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mL/kg
Arm/Group | rFVIIIFc 1000 IU | rFVIIIFc 3000 IU
Number analyzed (Participants) | 15 | 16
mL/kg | 52.59 [47.31 to 58.47] | 55.28 [47.12 to 64.84]

27. Secondary Outcome: Development of Inhibitor as Measured by the Nijmegen-Modified Bethesda Assay
Description: An inhibitor test result ≥0.6 Bethesda units (BU)/mL, confirmed on 2 separate samples drawn 2 to 4 weeks apart, was considered positive. Both tests were to be performed by the central laboratory using the Nijmegen-modified Bethesda Assay. An exact 95% confidence interval (CI) for the proportion of subjects with a confirmed inhibitor was calculated using the Clopper-Pearson method for a binomial proportion. Percentage of participants with confirmed inhibitor development was summarized overall.
Time Frame: Predose, Month 3, Month 6/early withdrawal. Additionally: If inhibitor suspected; at 10-15 EDs; 2-4 weeks prior to scheduled surgery; preoperatively on day of surgery; 1-2 weeks post-surgery; at last postoperative visit (last 2 for major surgery only)
Population: The Safety Analysis Set included participants who received at least 1 dose of rFVIIIFc.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- rFVIIIFc: Following the minimum 4-day washout, participants received their first injection of rFVIIIFc (on Injection 1 Day 1) rFVIIIFc 50 IU/kg at a strength of either 1000 or 3000 IU/vial. The second injection of rFVIIIFc 50 IU/kg at a strength of either 1000 or 3000 IU/vial was administered, in a crossover fashion, after a minimum of a 5-day washout (on Injection 2 Day 1).
  After completing the PK assessment, all participants began 1 of 3 continued treatment regimens for up to 6 months:
  1. A prophylaxis regimen at a starting dose of 50 IU/kg of rFVIIIFc given every 3 to 5 days; further dose and interval adjustments were based on the Investigator's discretion as needed to prevent or treat bleeding.
  2. A prophylaxis regimen of 65 IU/kg administered every 7 days was considered for appropriate participants who were selected based on the opinion of the Investigator.
  3. An episodic (on-demand) treatment with rFVIIIFc at 20 to 50 IU/kg, depending on the severity of the bleeding episode.
Arm/Group | rFVIIIFc
Number analyzed (Participants) | 19
percentage of participants | 0 [0 to 17.65]

ADVERSE EVENTS:
Time Frame: From screening (for serious adverse events) or first dose of study drug (for adverse events) until end of study (up to approximately 6 months).
Description: Adverse events presented are treatment-emergent (ie, those that occurred or worsened following the first injection of rFVIIIFc).
Groups:
- Total Active: Following the minimum 4-day washout, participants received their first injection of rFVIIIFc (on Injection 1 Day 1) rFVIIIFc 50 IU/kg at a strength of either 1000 or 3000 IU/vial. The second injection of rFVIIIFc 50 IU/kg at a strength of either 1000 or 3000 IU/vial was administered, in a crossover fashion, after a minimum of a 5-day washout (on Injection 2 Day 1).
  After completing the PK assessment, all participants began 1 of 3 continued treatment regimens for up to 6 months:
  1. A prophylaxis regimen at a starting dose of 50 IU/kg of rFVIIIFc given every 3 to 5 days; further dose and interval adjustments were based on the Investigator's discretion as needed to prevent or treat bleeding.
  2. A prophylaxis regimen of 65 IU/kg administered every 7 days was considered for appropriate participants who were selected based on the opinion of the Investigator.
  3. An episodic (on-demand) treatment with rFVIIIFc at 20 to 50 IU/kg, depending on the severity of the bleeding episode.
Arm/Group | Total Active
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 12/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Active (N=19)
Hydrocele (Congenital, familial and genetic disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Active (N=19)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 1
Post procedural cellulitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 2
Vitamin d deficiency (Metabolism and nutrition disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.